CLINICAL TRIAL: NCT06587646
Title: A Feasibility Study to Assess a "Virtual" (vEUA) Technology to Improve the Management of Perianal Crohn's Disease
Brief Title: VirtuAl Technology to Improve the Management of Perianal Crohn's (VAMP) - PROSPECTIVE
Acronym: VAMP-PROSPECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22CR004
Record Dates: First submitted 2024-09-02; First posted 2024-09-19 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Perianal Crohns Disease
Keywords: Perianal Crohn's Disease; 3D imaging; MRI

STUDY DESIGN:
Intervention Model Description: Patients randomised to either standard care or a virtual EUA (3D reconstruction imaging) via a computerised randomisation software.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (Active Comparator): Standard care (SC) will be defined as a written MRI report by a qualified radiologist followed by EUA and intervention as per surgeon's findings. Interventions will include one or combinations of: lay open of fistula, insertion of seton into the fistula tract and / or drainage of abscess. This arm is to provide outcome data on standard care for this condition as a comparator to the experimental arm.
  Interventions: Diagnostic Test: Standard Care - Written MRI report
- vEUA (Virtual Examination Under Anaesthetic) - 3D MRI imaging (Experimental): vEUA-enhanced care will be defined as having a vEUA performed by the radiologist following a MRI using the same unmodified sequence from the standard care (SC) arm (in addition to a written radiology report). The surgeon will then be given unlimited access to the vEUA interactive report via standard PC hardware. The surgeon will then perform the EUA and intervention as per SC but with the additional insight garnered from the vEUA interactive report. We will also monitor the time taken to mark up and produce the vEUA and compare this to the time taken to produce a standard MRI report.
  The care in this group will be the same as standard care but with the addition of 3D reconstruction of the MRI scan and review of this by the patient and surgeon.
  Interventions: Diagnostic Test: Virtual Examination under Anaeastehtic - 3D reconstruction imaging

INTERVENTIONS:
Diagnostic Test: Virtual Examination under Anaeastehtic - 3D reconstruction imaging — 3D reconstruction of MRI imaging and review by patient and surgeon prior to surgical intervention.
  Arms: vEUA (Virtual Examination Under Anaesthetic) - 3D MRI imaging
Diagnostic Test: Standard Care - Written MRI report — A standard written MRI report will be provided to the surgeon and patient prior to surgical intervention.
  Arms: Standard Care

SUMMARY:
Crohn's is an inflammatory condition that can affect any part of the gut. Over half a million people in the UK live with Crohn's disease and about a quarter will develop a fistula near their back passage. A fistula is an abnormal connection between two surfaces of the body. These can be hard to treat causing pain and infection. Surgery is required to control infection and in extreme cases this can lead to incontinence or even formation of a stoma, when the bowel is brought to the skin and waste goes into a bag on the tummy wall.

Patients with perianal Crohn's are usually referred to a surgeon by their medical team and subsequently undergo a MRI scan and an examination under anaesthesia (EUA) where abscesses (regions of fluid build-up) will be drained and a seton (plastic sling or suture) inserted through the fistula, or the fistula opened to the skin if this will not affect continence. They are then started on specialist medication by the gastroenterologists (gut doctors).

Abscesses or fistulas can be difficult to identify during EUA, leading to ongoing infection and repeat procedures. This causes additional scarring and delays the medical treatment that can allow fistulas to heal. Multiple or incorrectly performed operations can also damage the muscles that help hold stool in the back passage, leading to incontinence.

We believe that improving how information is communicated between radiology (who report scans) and surgeons will improve their ability to identify and manage all fistulas and collections at operation. Here is a typical MRI report given to the surgeon by the radiologist:

'There is a low intersphincteric fistula with predicted internal opening in the lower half of the anal canal at dentate line level between 5-6 o'clock that passes in the intersphincteric plane to the anal verge between 5-6 o'clock.'

This protocol was developed in an era when written communication was really the only way to convey information between specialists. Jargon aside, surgeons face significant difficulty interpreting such written descriptions of a complex 3D structure and using it as a surgical guide. Indeed, a major complaint from surgeons is how difficult it is to get real value from these preoperative MRIs, which cost time and money.

With advances in digital technology, we believe this system can be vastly improved.

Motilent (a UK SME specialising in technology to improve the management of Crohn's Disease) has developed a sophisticated visualisation tool to provide a 3D model of the fistula and surrounding structures, we call this tool Virtual EUA (vEUA), allowing the surgeon to better understand the anatomy of the problem in conjunction with radiology.

We are aiming to establish whether vEUA changes the behaviour of colorectal surgeons, increasing confidence in identifying and dealing with fistulas, which will reduce the number of surgical procedures required and improve the quality of care, resulting in a cost saving for the hospital and a much-needed step towards more effective management of perianal Crohn's.

Any patient taking part in the trial will be randomly allocated to have the 3D model utilised in their care or standard care. We will use pre- and post-surgical patient questionnaires, surgical questionnaires and MRI imaging to establish if vEUA is safe and effective in improving the care of patients with perianal Crohn's.

DETAILED DESCRIPTION:
The development of the vEUA tool is a significant advancement in the management of perianal Crohn's disease fistulas. Mismanagement of fistulas can lead to significant complications, such as abscesses, scarring, and delayed healing. Additionally, multiple surgeries can cause damage to the anal sphincter muscles, leading to incontinence and other issues.

With the vEUA tool, surgeons can now have a more precise and accurate understanding of the fistula anatomy before conducting the examination under anaesthesia. This approach can significantly reduce the risk of misdiagnosis and subsequent complications. The tools 3D visualization capability allows surgeons to assess the extent of the fistula, its location, and any associated abscesses or inflammation. This information is essential for planning the surgery and ensuring that the procedure is as minimally invasive as possible.

In addition to improving surgical planning, the vEUA tool can also enhance post-operative care. The 3D model generated by the tool can be used to monitor the healing process and ensure that the fistula has healed correctly. This approach reduces the need for multiple follow-up surgeries and promotes faster healing. With the vEUA tool, surgeons can better plan the surgery to avoid damaging the muscles, promoting faster healing and reducing the risk of long-term complications.

Overall, the development of the vEUA tool represents a significant breakthrough in the management of Crohn's disease and perianal fistulas. The tool's ability to provide a more precise and accurate understanding of the fistula's anatomy will reduce the risk of misdiagnosis, promote faster healing, and improve patient outcomes.

vEUA generates a disease activity score based on T2 enhancement and a volumetric measurement of the fistula tract, providing a more detailed analysis of the fistula and surrounding structures.

RESEARCH QUESTION / AIM(S) Our proposed investigation aims to generate early clinical usage data to assess the feasibility of the vEUA approach. Our findings will feed into a larger multicentre study at a later date.

In this early-stage investigation, we aim to answer the question:

Does vEUA improve the surgeon's confidence in and ability to manage all fistula tracts and drain all collections in perianal Crohn's disease at surgery?

In addition, we aim to gain insight into the following supplementary questions that will feed into future projects:

* Can vEUA be used effectively by trained radiologists?
* How long does it take a radiologist to perform a vEUA?
* What concerns do patients have over the vEUA system? How does viewing a vEUA report change their perception of their disease, their treatment and their ability to provide informed consent? (Answered through our PPIE work packages and survey).
* Is there any indication that the vEUA system reduces the likelihood of a patient requiring multiple operations to control sepsis and fistula tracts?
* Does the use of vEUA translate to improved disease control and a subsequent improvement in quality of life for patients?

The purpose of answering these questions is to determine whether the quality of care afforded to perianal Crohn's patients can be meaningfully improved by the vEUA system. These data will highlight which patients will benefit most from vEUA. It is possible that this technology will be most useful for those with more complex disease, i.e., multiple fistula tracts or deep collections, thus ensuring value for money in the future through correct patient selection to vEUA.

30 patients will be prospectively recruited to this vEUA feasibility study, 15 to standard care and 15 randomised to the vEUA technology, and assess outcome data as outlined below to guide future studies and assess the acceptability of the vEUA technology to patients and clinicians.

Standard care (SC) will be defined as a written MRI report by a qualified radiologist followed by EUA and intervention as per surgeon's findings. Interventions will include one or combinations of: lay open of fistula, insertion of seton into the fistula tract and / or drainage of abscess.

vEUA-enhanced care will be defined as having a vEUA performed by the radiologist following a MRI using the same unmodified sequence from the SC arm (in addition to a written radiology report). The surgeon will then be given unlimited access to the vEUA interactive report via standard PC hardware. The surgeon will then perform the EUA and intervention as per SC but with the additional insight garnered from the vEUA interactive report. We will also monitor the time taken to mark up and produce the vEUA and compare this to the time taken to produce a standard MRI report.

OUTCOME MEASURES:

These will include:

1. Baseline inflammatory bowel disease (IBD) specific patient outcome measures will be collected on recruitment, including:

   * IBD quality of life (IBDQ) scores
   * The Crohn's Anal Fistula Quality of Life (CAF-QoL) scale
   * Hospital Anxiety and Depression Scale (HADS)
   * Incontinence (Vaizey / St. Marks) score
2. Baseline clinical outcome measures will be assessed including:

   * Perianal Disease Activity Score (PDAI)
   * Number of surgical interventions (EUAs) in previous 3 months
   * Number of antibiotic courses in previous 3 months
3. Biochemical disease activity will be measured by:

   * C-reactive protein (CRP)
   * Faecal calprotectin These outcome measures will be re-captured again at 3 months postoperatively and exploratory analyses will be undertaken. We will use baseline variables to predict postoperative response.
4. An evaluation of surgical confidence and opinion will be used to assess surgical confidence prior to commencement of the procedure, surgeons will be asked to propose and document a likely pre-operative plan based on their understanding of the anatomy of the disease from the information available through either a standard MRI report or vEUA. Their confidence in this plan will be scored using a Likert scale from 1 (no confidence) to 10 (extremely confident). Immediately following surgery, surgeons will again be asked to complete a questionnaire to include interventions completed, adherence to pre-operative plan scored from 1 (no adherence to plan) to 10 (exact plan followed) and their confidence in having adequately and safely identified and treated all fistula and collections with each aspect scored from 1 (no confidence) to 10 (extremely confident).
5. An evaluation of patient opinion will help us understand the benefit of vEUA in describing and explaining disease anatomy to the patient and in obtaining informed consent for surgical intervention. Patients will be presented with a decisional conflict scale10 to evaluate their personal uncertainty related to their surgery after consultation with a surgeon. A 16-question, 5-response category (strongly disagree to strongly agree) traditional decisional conflict scale will be to assess whether the patient feels they are making an effective decision (i.e., the decision is informed, values-based and likely to be implemented). Results will be compared between patients shown their vEUA and those randomised to SC.
6. A radiological assessment of surgical quality will allow assessment of disease control at surgery. Patients will undergo a repeat MRI scan of the pelvis at 4 weeks post-procedure to look for undrained collections, the size of any remaining collections or untreated fistula i.e., those not laid open or with a seton in-situ. MRI scans will be reviewed by an adjudication radiology / surgical panel to compare the relative successes of SC and vEUA in achieving disease control.

We hope to establish utilising these data that vEUA is safe and effective in improving the care of patients with perianal Crohn's.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent
* Active perianal Crohn's disease as defined by clinical assessment with fistula or abscess formation
* A clinical decision has been taken that surgery is required for perianal disease
* Ages of 18-75

Exclusion Criteria:

* Inability to consent
* history of Proctectomy,
* absence of a diagnosis of Crohn's disease,
* perianal fistulising disease not secondary to Crohn's disease,
* Rectovaginal fistulas
* Malignant disease
* Significant cardiovascular or respiratory disease
* Neurological or cognitive impairment
* Significant physical disability
* Significant hepatic disease or renal failure
* Subjects currently (or in the last three months) participating in another research project
* Pregnancy or breastfeeding
* If MRI is contraindicated (e.g. pacemaker).
* under 18 years old or over 75 years old

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2026-07-23 (Estimated); Study Completion 2026-09-07 (Estimated)

PRIMARY OUTCOMES:
Clinical disease activity assessment | Enrollment to 3 months post-intervention
  Clinical outcome measures will be assessed by Perianal Disease Activity Score (PDAI)
Clinical disease activity assessment | Enrollment to 3 months post-intervention
  Clinical outcome measures will be assessed by number of surgical interventions (EUAs) in previous 3 months
Clinical disease activity assessment | Enrollment to 3 months post-intervention
  Clinical outcome measures will be assessed by number of antibiotic courses in previous 3 months
Patient reported outcomes | Enrollment to 3 months post-intervention
  Inflammatory bowel disease (IBD) specific patient outcome measures will be collected on recruitment and after intervention using The Crohn's Anal Fistula Quality of Life (CAF-QoL) scale
Patient reported outcomes | Enrollment to 3 months post-intervention
  Inflammatory bowel disease (IBD) specific patient outcome measures will be collected on recruitment and after intervention using Hospital Anxiety and Depression Scale (HADS)
Patient reported outcomes | Enrollment to 3 months post-intervention
  Inflammatory bowel disease (IBD) specific patient outcome measures will be collected on recruitment and after intervention using IBD quality of life (IBDQ) scores
Patient reported outcomes | Enrollment to 3 months post-intervention
  Inflammatory bowel disease (IBD) specific patient outcome measures will be collected on recruitment and after intervention using Incontinence (Vaizey / St. Marks) score
Biochemical disease activity monitoring | Enrollment to 3 months post-intervention
  Biochemical disease activity will be measured byC-reactive protein (CRP)
Biochemical disease activity monitoring | Enrollment to 3 months post-intervention
  Biochemical disease activity will be measured by Faecal calprotectin
Disease control at surgery / surgical success | 4-8 weeks post-surgery
  To assess disease control at surgery patients will undergo a repeat MRI scan of the pelvis at 4-8 weeks post-procedure to look for undrained collections
Disease control at surgery / surgical success | 4-8 weeks post-surgery
  To assess disease control at surgery patients will undergo a repeat MRI scan of the pelvis at 4-8 weeks post-procedure to look at the size of any remaining collections or untreated fistula i.e. those not laid open or with a seton in-situ
Disease control at surgery / surgical success | 4-8 weeks post-surgery
  To assess disease control at surgery patients will undergo a repeat MRI scan and MRI scans will be reviewed by an adjudication radiology / surgical panel to compare the relative successes of standard care and vEUA in achieving disease control.
Clinical disease activity assessment | Enrollment to 3 months post-intervention
  Clinical outcome measures will be assessed using Perianal Disease Activity Score (PDAI)
Clinical disease activity assessment | Enrollment to 3 months post-intervention
  Clinical outcome measures will be assessed using Number of surgical interventions (EUAs) in previous 3 months
Clinical disease activity assessment | Enrollment to 3 months post-intervention
  Clinical outcome measures will be assessed using Number of antibiotic courses in previous 3 months

SECONDARY OUTCOMES:
Evaluation of surgical confidence and opinion data | up to 4 weeks pre and up to 4 weeks post-surgical intervention
  To assess surgical confidence prior to commencement of the procedure, surgeons will be asked to propose and document a likely pre-operative plan based on their understanding of the anatomy of the disease from the information available through either a standard MRI report or vEUA. Their confidence in this plan will be scored using a Likert scale from 1 (no confidence) to 10 (extremely confident). Immediately following surgery, surgeons will again be asked to complete a questionnaire to include interventions completed, adherence to pre-operative plan scored from 1 (no adherence to plan) to 10 (exact plan followed) and their confidence in having adequately and safely identified and treated all fistula and collections with each aspect scored from 1 (no confidence) to 10 (extremely confident).

CONTACTS AND LOCATIONS:
Locations (1):
- Nottingham University Hospital NHS Trust, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Will be for publication rather than data sharing